CLINICAL TRIAL: NCT06555432
Title: Post-Marketing Surveillance (Usage Results Study) of LIVTENCITY Tablet (Maribavir) for the Approved Indications in South Korea
Brief Title: A Study of LIVTENCITY (Maribavir) in Adults With Cytomegalovirus (CMV) Infection After Transplantation in South Korea
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-620-4002
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cytomegalovirus (CMV)
Keywords: Drug Therapy
MeSH Terms: interventions — maribavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- All Participants: Participants with post-transplant CMV infection and/or disease who are refractory and/or resistant to one or more prior therapy (including ganciclovir, valganciclovir, foscarnet or cidofovir) will be treated with LIVTENCITY tablet as per treating physician's discretion in a routine clinical practice setting, according to the approved labelling and will be observed prospectively for up to a 20-week period.
  Interventions: Drug: LIVTENCITY

INTERVENTIONS:
Drug: LIVTENCITY — LIVTENCITY tablet.
  Other Names: Maribavir

SUMMARY:
Cytomegalovirus (CMV) is a common virus that infects many people. It can cause serious illness in people with weak immune systems especially in those undergoing transplants. LIVTENCITY (Maribavir) is a medicine approved for treating CMV infection in adults after transplant in South Korea.

The main aim of this study is to learn how safe and effective LIVTENCITY (Maribavir) is in treating adults with CMV infection after transplant in a routine clinical practice setting.

During the study, a participant's data will be collected for about 5 months (20 weeks). The study does not have fixed visits to the hospital, but it is recommended to visit the study doctor approximately 6 times during study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with post-transplant CMV infection and/or disease who are refractory and/or resistant to one or more prior therapy including ganciclovir, valganciclovir, cidofovir or foscarnet.
* Participants with age greater than or equal to (>=) 19 years.
* Initiate first treatment course with maribavir.
* Voluntarily consent to participate in the study.

Exclusion Criteria:

* Participants for whom LIVTENCITY Tablet (maribavir) is contraindicated as per product label.
* Participants previously treated with maribavir in any study or as marketed drug.
* Participants actively participating in other clinical trials of post-transplant CMV infection treatment or with other experimental treatments.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with post-transplant CMV infection and/or disease who are refractory and/or resistant to one or more prior therapy including ganciclovir, valganciclovir, foscarnet or cidofovir and initiate maribavir treatment for the first time will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs), Causality to AEs, Serious AEs (SAEs) and AEs of Special Interest (AESI) | Up to Week 20
  Number of participants with AEs, causality to AEs, SAEs and AESI will be reported. The investigator will assess the causal relationship (causality) between the medicinal product and the AE using his/her clinical expertise and judgment.
Number of Participants With Expected/Unexpected AEs and SAEs | Up to Week 20
  Unexpected AE is defined as AE that differs from the information in the product label in nature, severity, specificity, or outcome.
Number of Participants With Adverse Drug Reactions (ADRs), Unexpected ADRs, Expected ADRs, Serious ADRs (SADRs) Expected SADRs and Unexpected SADRs | Up to Week 20
  An ADR refers to a harmful and unintended reaction that occurs when an investigational product is normally administered or used, and when the causal relationship between the reaction and the investigational product cannot be ruled out. Among voluntarily reported AEs, if the causality between the AE and the investigational product is not known, it is considered an ADR. However, if both the reporter and the manufacturer/sponsor determine that the case is unrelated to the investigational product, it is excluded from being classified as an ADR. Serious ADR means noxious or unintended response to a drug that occurs at any dosage and that requires in-patient hospitalization or prolongation of existing hospitalization, causes congenital malformation, results in persistent or significant disability or incapacity, is life-threatening or results in death. Unexpected ADRs is defined as ADR that differs from the information in the product label in nature, severity, specificity, or outcome.
Number of Participants With Special Situation Report (SSR) | Up to Week 20
  SSR include following events: Pregnancy: any case in which a pregnancy participant is exposed to a Takeda Product or in which a female participant or partner of a male participant becomes pregnant following Takeda product.; Breastfeeding: infant exposure from breast milk; Overdose: all information of any accidental or intentional overdose; Drug abuse, misuse or medication error: all information on medicinal product (MP) abuse, misuse of medication error (potential or actual); Suspected transmission of infectious agent: Suspected (in sense of confirmed or potential) transmission of infectious agent by a MP; Lack of efficacy of Takeda Product; accidental/occupational exposure; Use outside the terms of the marketing authorization, also known as "off-label" and "off-label use" for unintended benefit; Use of falsified and counterfeit MP; Drug-drug and drug-food interactions; Inadvertent or accidental exposure with or without an AE; AEs occurring in the pediatric or elderly population.

SECONDARY OUTCOMES:
Percentage of Participants With CMV Viremia Clearance as Assessed by Polymerase Chain Reaction (PCR) | At Weeks 2, 8 and the last dose (up to 20 weeks)
  CMV viremia clearance will be defined as CMV deoxyribonucleic acid (DNA) concentration below the lower limit of quantification (<LLOQ) or predefined threshold of each device. The assessment will be done using PCR.
Percentage of Participants Who Achieved CMV Infection Symptom Control | At Weeks 2, 8 and the last dose (up to 20 weeks)
  CMV infection symptom control will be defined as resolution or improvement of tissue invasive CMV disease or CMV syndrome for participants symptomatic at baseline or no symptoms of tissue invasive CMV disease or CMV syndrome for subjects asymptomatic at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/8b425af2ffa2462a??page=1&idFilter=TAK-620-4002